CLINICAL TRIAL: NCT01851512
Title: Single-Blind, Randomized, Comparative, Phase I Study to Evaluate the Tolerability, Safety, and Pharmacokinetic Characteristics of Human Chorionic Gonadotropin Between Two Recombinant hCG Products, DA-3803 Injection and Ovidrel Liquid Injection, in Healthy Subjects
Brief Title: A Study to Evaluate the Tolerability, Safety and Pharmacokinetic Characteristics of DA-3803
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Dong-A ST Co., Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DA3803_HCG_I
Record Dates: First submitted 2013-05-08; First posted 2013-05-10 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Infertility; Induction of Ovulation
MeSH Terms: conditions — Infertility | interventions — Drug Evaluation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- T-R (Test-Reference drug) (Experimental): DA-3803 Injection is injected first and Ovidrel liquid injection is injected after 3-week period
  Interventions: Drug: T-R (Test-Reference drug)
- R-T (Reference-Test drug) (Experimental): Ovidrel liquid injection is injected first and DA-3803 Injection is injected after 3-week period
  Interventions: Drug: R-T (Reference-Test drug)

INTERVENTIONS:
Drug: T-R (Test-Reference drug)
  Other Names: Drug: DA-3803 (Test drug); Drug: Ovidrel liquid injection (Referecne drug)
  Arms: T-R (Test-Reference drug)
Drug: R-T (Reference-Test drug)
  Other Names: Drug: Ovidrel liquid injection (Referecne drug); Drug: DA-3803 (Test drug)
  Arms: R-T (Reference-Test drug)

SUMMARY:
This is a single-blind, randomized, comparative, phase I study to evaluate the tolerability, safety and pharmacokinetic characteristics of human chorionic gonadotropin between two recombinant hCG products named DA-3803 injection and ovidrel liquid injection, in healthy subjects. The subjects will injected with these two injections at the the 21day-interval of time and their conditions including vital signs, blood, clinical examination will be carefully observed.

ELIGIBILITY:
Inclusion Criteria:

* No medical history relating to the alimentary system, liver system, heart system, haematological disease
* Ideal body weight +/- 20%

Exclusion Criteria:

* acute disease within 28 days
* medical history that might affect the absorption, distribution, secretion, metabolism of drugs
* metrectomy surgery
* desexualization
* tubal ligation
* menopause
* pregnancy
* not able to use contraception
* drink alcohol more than 14 units/week
* smoker who smokes 10 or more cigarettes

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2010-05; Primary Completion 2010-08 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Concentration in serum of hCG examined by non-compartmental analysis | 3 weeks
  Examine the following:
  * Maximum blood concentration
  * Travel time of maximum blood concentration
  * half time t(1/2)
  * Clearance
  * Volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Young Park, M.D., Ph.D., Principal Investigator — Korea University Anam Hospital; Kyoung-Ah Kim, Ph.D., Study Director — Korea University Anam Hospital; Un Jip Kim, M.D., Ph.D., Study Director — Korea University Anam Hospital; Soo Kyung Kim, M.D., Ph.D., Study Director — Korea University Anam Hospital; Hyun Tae Park, M.D., Ph.D., Study Director — Korea University Anam Hospital